CLINICAL TRIAL: NCT00032162
Title: Phase I/II Trial, Dose Finding Combination Chemotherapy With PegLiposomal Doxorubicin (PLD) And Carboplatin In Patients With Gynecologic Tumors
Brief Title: Liposomal Doxorubicin and Carboplatin in Treating Patients With Gynecologic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AGO Study Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069262; AGOSG-AGO-GYN-2; EU-20147
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Cervical Cancer; Endometrial Cancer; Fallopian Tube Cancer; Ovarian Cancer; Sarcoma
Keywords: stage III cervical cancer; recurrent cervical cancer; stage IB cervical cancer; stage IIB cervical cancer; stage IVB cervical cancer; stage IA cervical cancer; stage IIA cervical cancer; stage IVA cervical cancer; stage I endometrial carcinoma; stage II endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma; recurrent endometrial carcinoma; fallopian tube cancer; stage I uterine sarcoma; stage II uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma; ovarian sarcoma; ovarian carcinosarcoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Sarcoma | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PLD (Experimental): dose finding study of PLD in combination with Carboplatin
  Interventions: Drug: carboplatin; Drug: pegylated liposomal doxorubicin hydrochloride

INTERVENTIONS:
Drug: carboplatin — AUC 6 q4w
Drug: pegylated liposomal doxorubicin hydrochloride — 20/30/40 mg/qm q4w Dose finding study

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining liposomal doxorubicin with carboplatin in treating patients who have gynecologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of doxorubicin HCl liposome when administered with carboplatin in patients with gynecological tumors.
* Determine the dose-limiting toxicity of this regimen in these patients.
* Determine the kind, frequency, severity, and duration of adverse events in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of doxorubicin HCl liposome.

Patients receive doxorubicin HCl liposome IV over 60 minutes followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 28 days for 6 courses.

Cohorts of 3-6 patients receive escalating doses of doxorubicin HCl liposome until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued and treated at the MTD as above.

Patients are followed at 4-6 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 12-24 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed fallopian tube cancer, Muellerian mixed tumor, endometrial cancer, uterine sarcoma, ovarian cancer with sarcoma parts, or cervical cancer

  * No ovarian epithelial cancer

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 70-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin greater than 10.0 g/dL

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal

Renal:

* Glomerular filtration rate at least 60 mL/min

Cardiovascular:

* No atrial or ventricular arrhythmias
* No congestive heart failure even if stabilized on medication
* No New York Heart Association class III or IV heart disease
* No myocardial infarction within the past 6 months

Other:

* No pre-existing sensory or motor neuropathy grade 2 or greater
* No active infection
* No other serious medical condition that would preclude study
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy

Chemotherapy:

* No more than 1 prior chemotherapy regimen for the malignancy
* No other concurrent chemotherapy

Endocrine therapy:

* Prior hormonal therapy within the past 10 days allowed
* No concurrent hormonal therapy

Radiotherapy:

* At least 6 weeks since prior radiotherapy to no more than 25% of bone marrow

Surgery:

* Not specified

Other:

* At least 30 days since prior experimental agents
* No other concurrent therapies that would preclude study
* No concurrent participation in another study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2001-08; Primary Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
DL DLT | DLT during first 3 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Andreas du Bois, MD, PhD, Study Chair — Dr. Horst-Schmidt-Kliniken
Locations (19):
- Germany (19):
  - Universitaetsklinikum Charite, Berlin
  - Zentralkrankenhaus, Bremen
  - Medizinische Klinik I, Dresden
  - Universitaetsklinik Duesseldorf, Düsseldorf
  - Evangelisches Krankenhaus, Düsseldorf
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Staedtisches Krankenhaus FFM-Hoechst, Frankfurt am Main
  - Universitaetsklinik Goettingen, Göttingen
  - Klinik Fuer Innere Medizin Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Frauenklinik der MHH, Hanover
  - Vincentius Krankenhaus, Karlsruhe
  - Christian-Albrechts University of Kiel, Kiel
  - Klinik der Otto - v. - Guericke - Universitat, Magdeburg
  - Klinikum Grosshadern, Munich (Muenchen)
  - Klinikum Rechts Der Isar/Technische Universitaet Muenchen, Munich (Muenchen)
  - Klinik und Poliklinik fuer Kinderheilkunde, Münster
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaet Ulm, Ulm
  - Dr. Hors t- Schmidt - Kliniken, Wiesbaden

REFERENCES:
- [Result] du Bois A, Pfisterer J, Burchardi N, Loibl S, Huober J, Wimberger P, Burges A, Stahle A, Jackisch C, Kolbl H; Arbeitsgemeinschaft Gynaekologische Onkologie Studiengruppe Ovarialkarzinom; Kommission Uterus. Combination therapy with pegylated liposomal doxorubicin and carboplatin in gynecologic malignancies: a prospective phase II study of the Arbeitsgemeinschaft Gynaekologische Onkologie Studiengruppe Ovarialkarzinom (AGO-OVAR) and Kommission Uterus (AGO-K-Ut). Gynecol Oncol. 2007 Dec;107(3):518-25. doi: 10.1016/j.ygyno.2007.08.008. Epub 2007 Oct 25. PMID 17910981